CLINICAL TRIAL: NCT02978157
Title: A Prospective Randomized Trial of Levofloxacin-amoxicillin Triple Therapy vs. Levofloxacin-tetracycline Quadruple Therapy in Second-line Helicobacter Pylori Treatment
Brief Title: Levofloxacin Triple and Bismuth Quadruple Therapies for Rescue Treatment of H Pylori Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Collaborators: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Principal Investigator, Ping-I (William) Hsu, M.D., Professor, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VGHKS104-062
Record Dates: First submitted 2016-11-28; First posted 2016-11-30 (Estimated); Results first posted 2019-03-14 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; Eradication rate; Rescue treatment
MeSH Terms: interventions — Esomeprazole; Amoxicillin; Levofloxacin; Bismuth; Tetracycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- esomeprazole+amox+levo (Active Comparator): esomeprazole 40 mg b.d., amoxicillin 500 mg q.d.s., and levofloxacin 500 mg o.d.
  Interventions: Drug: esomeprazole+amox+levo
- esomeprazole+bismuth+tetra+levo (Experimental): esomeprazole 40 mg b.d., bismuth 120 mg q.d.s., tetracycline 500 mg q.d.s., and levofloxacin 500 mg o.d.
  Interventions: Drug: esomeprazole+bismuth+tetra+levo

INTERVENTIONS:
Drug: esomeprazole+amox+levo — esomeprazole 40 mg b.d., amoxicillin 500 mg q.d.s., levofloxacin 500 mg o.d.
  Other Names: esomeprazole 40 mg; amoxicillin 500 mg; levofloxacin 500 mg
  Arms: esomeprazole+amox+levo
Drug: esomeprazole+bismuth+tetra+levo — esomeprazole 40 mg b.d., bismuth 120 mg q.d.s., tetracycline 500 mg q.d.s., and levofloxacin 500 mg o.d.
  Other Names: esomeprazole 40mg; bismuth 120 mg; tetracycline 500 mg; levofloxacin 500 mg
  Arms: esomeprazole+bismuth+tetra+levo

SUMMARY:
From the profiles of antibiotic susceptibility data following eradication therapy, tetracycline, amoxicillin and levofloxacin are all good candidates of antibiotics used in the rescue treatment.

DETAILED DESCRIPTION:
The H pylori-infected adult patients with failure of standard triple therapy and H pylori-infected adult patients with failure of non-bismuth quadruple therapy are randomly assigned to either EAL (esomeprazole 40 mg b.d., amoxicillin 500 mg q.d.s., and levofloxacin 500 mg o.d.) or EBTL (esomeprazole 40 mg b.d., bismuth 500 mg q.d.s., tetracycline 500 mg q.d.s., and levofloxacin 500 mg o.d.) therapy for 10 days. Repeated endoscopy with rapid urease test, histological examination and culture or urea breath tests is performed at six weeks after the end of anti-H pylori therapy.

ELIGIBILITY:
Inclusion Criteria:

* positive results of both rapid urease test and histology,
* a positive result of urea breath test,
* or a positive result of culture.

Exclusion Criteria:

* ingestion of antibiotics, bismuth, or proton pump inhibitor（PPI）within the prior 4 weeks,
* patients with allergic history to the medications used,
* patients with previous gastric surgery,
* the coexistence of serious concomitant illness (for example, decompensated liver cirrhosis, uremia),
* pregnant women

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2015-02; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ping-I Hsu, Study Chair — Kaohsiung Veterans General Hospital.
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Suerbaum S, Michetti P. Helicobacter pylori infection. N Engl J Med. 2002 Oct 10;347(15):1175-86. doi: 10.1056/NEJMra020542. No abstract available. PMID 12374879
- [Background] Zucca E, Dreyling M; ESMO Guidelines Working Group. Gastric marginal zone lymphoma of MALT type: ESMO clinical recommendations for diagnosis, treatment and follow-up. Ann Oncol. 2009 May;20 Suppl 4:113-4. doi: 10.1093/annonc/mdp146. No abstract available. PMID 19454427
- [Background] Asaka M, Kato M, Takahashi S, Fukuda Y, Sugiyama T, Ota H, Uemura N, Murakami K, Satoh K, Sugano K; Japanese Society for Helicobacter Research. Guidelines for the management of Helicobacter pylori infection in Japan: 2009 revised edition. Helicobacter. 2010 Feb;15(1):1-20. doi: 10.1111/j.1523-5378.2009.00738.x. PMID 20302585
- [Background] Fock KM, Katelaris P, Sugano K, Ang TL, Hunt R, Talley NJ, Lam SK, Xiao SD, Tan HJ, Wu CY, Jung HC, Hoang BH, Kachintorn U, Goh KL, Chiba T, Rani AA; Second Asia-Pacific Conference. Second Asia-Pacific Consensus Guidelines for Helicobacter pylori infection. J Gastroenterol Hepatol. 2009 Oct;24(10):1587-600. doi: 10.1111/j.1440-1746.2009.05982.x. PMID 19788600
- [Background] Graham DY, Fischbach L. Helicobacter pylori treatment in the era of increasing antibiotic resistance. Gut. 2010 Aug;59(8):1143-53. doi: 10.1136/gut.2009.192757. Epub 2010 Jun 4. PMID 20525969
- [Background] Gumurdulu Y, Serin E, Ozer B, Kayaselcuk F, Ozsahin K, Cosar AM, Gursoy M, Gur G, Yilmaz U, Boyacioglu S. Low eradication rate of Helicobacter pylori with triple 7-14 days and quadriple therapy in Turkey. World J Gastroenterol. 2004 Mar 1;10(5):668-71. doi: 10.3748/wjg.v10.i5.668. PMID 14991935
- [Background] Gatta L, Vakil N, Leandro G, Di Mario F, Vaira D. Sequential therapy or triple therapy for Helicobacter pylori infection: systematic review and meta-analysis of randomized controlled trials in adults and children. Am J Gastroenterol. 2009 Dec;104(12):3069-79; quiz 1080. doi: 10.1038/ajg.2009.555. Epub 2009 Oct 20. PMID 19844205
- [Background] Wu DC, Hsu PI, Wu JY, Opekun AR, Kuo CH, Wu IC, Wang SS, Chen A, Hung WC, Graham DY. Sequential and concomitant therapy with four drugs is equally effective for eradication of H pylori infection. Clin Gastroenterol Hepatol. 2010 Jan;8(1):36-41.e1. doi: 10.1016/j.cgh.2009.09.030. Epub 2009 Oct 3. PMID 19804842
- [Background] Malfertheiner P, Megraud F, O'Morain CA, Atherton J, Axon AT, Bazzoli F, Gensini GF, Gisbert JP, Graham DY, Rokkas T, El-Omar EM, Kuipers EJ; European Helicobacter Study Group. Management of Helicobacter pylori infection--the Maastricht IV/ Florence Consensus Report. Gut. 2012 May;61(5):646-64. doi: 10.1136/gutjnl-2012-302084. PMID 22491499
- [Background] Hojo M, Miwa H, Nagahara A, Sato N. Pooled analysis on the efficacy of the second-line treatment regimens for Helicobacter pylori infection. Scand J Gastroenterol. 2001 Jul;36(7):690-700. doi: 10.1080/003655201300191941. PMID 11444467
- [Background] Saad RJ, Schoenfeld P, Kim HM, Chey WD. Levofloxacin-based triple therapy versus bismuth-based quadruple therapy for persistent Helicobacter pylori infection: a meta-analysis. Am J Gastroenterol. 2006 Mar;101(3):488-96. doi: 10.1111/j.1572-0241.2006.00637.x. PMID 16542284
- [Background] Pontone S, Standoli M, Angelini R, Pontone P. Efficacy of H. pylori eradication with a sequential regimen followed by rescue therapy in clinical practice. Dig Liver Dis. 2010 Aug;42(8):541-3. doi: 10.1016/j.dld.2009.12.007. Epub 2010 Jan 12. PMID 20061196
- [Background] Gisbert JP, Molina-Infante J, Marin AC, Vinagre G, Barrio J, McNicholl AG. Second-line rescue triple therapy with levofloxacin after failure of non-bismuth quadruple "sequential" or "concomitant" treatment to eradicate H. pylori infection. Scand J Gastroenterol. 2013 Jun;48(6):652-6. doi: 10.3109/00365521.2013.786132. Epub 2013 Apr 5. PMID 23556551
- [Background] Hsu PI, Lai KH, Tseng HH, Liu YC, Yen MY, Lin CK, Lo GH, Huang RL, Huang JS, Cheng JS, Huang WK, Ger LP, Chen W, Hsu PN. Correlation of serum immunoglobulin G Helicobacter pylori antibody titers with histologic and endoscopic findings in patients with dyspepsia. J Clin Gastroenterol. 1997 Dec;25(4):587-91. doi: 10.1097/00004836-199712000-00007. PMID 9451668
- [Background] Peng NJ, Lai KH, Liu RS, Lee SC, Tsay DG, Lo CC, Tseng HH, Huang WK, Lo GH, Hsu PI. Endoscopic 13C-urea breath test for the diagnosis of Helicobacter pylori infection. Dig Liver Dis. 2003 Feb;35(2):73-7. doi: 10.1016/s1590-8658(03)00014-8. PMID 12747623
- [Background] Peng NJ, Lai KH, Liu RS, Lee SC, Tsay DG, Lo CC, Tseng HH, Huang WK, Lo GH, Hsu PI. Clinical significance of oral urease in diagnosis of Helicobacter pylori infection by [13C]urea breath test. Dig Dis Sci. 2001 Aug;46(8):1772-8. doi: 10.1023/a:1010626225949. PMID 11508681
- [Background] Kita T, Sakaeda T, Aoyama N, Sakai T, Kawahara Y, Kasuga M, Okumura K. Optimal dose of omeprazole for CYP2C19 extensive metabolizers in anti-Helicobacter pylori therapy: pharmacokinetic considerations. Biol Pharm Bull. 2002 Jul;25(7):923-7. doi: 10.1248/bpb.25.923. PMID 12132671

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1. recruitment period: February 2015
  2. Type of location: Kaohsiung Veterans General Hospital and Kaohsiung Medical University Chung-Ho Memorial Hospital
Pre-assignment Details: None were excluded following participant enrollment.
Period: Overall Study
Arm/Group | Esomeprazole+Amox+Levo | Esomeprazole+Bismuth+Tetra+Levo
Started | 52 | 50
Completed | 52 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients received levoflaxacin triple therapy
Groups:
- Total: Total of all reporting groups
Arm/Group | Esomeprazole+Amox+Levo | Esomeprazole+Bismuth+Tetra+Levo | Total
Number analyzed (Participants) | 52 | 50 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 39 | 40 | 79
  >=65 years | 13 | 10 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.08 (13.55) | 56.38 (12.81) | 55.72 (13.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 25 | 60
  Male | 17 | 25 | 42
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 52 | 50 | 102
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Taiwan | 52 | 50 | 102
history of smoking [Number; unit: participants] | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants in Which H. Pylori Was Eradicated
Description: Number of participants with negative H pylori status in follow-up tests as a measure of successful eradication
Time Frame: six weeks after the end of anti-H pylori therapy.
Population: Intention to treat
Measure: Number; unit: participants
Arm/Group | Esomeprazole+Amox+Levo | Esomeprazole+Bismuth+Tetra+Levo
Number analyzed (Participants) | 52 | 50
participants | 36 | 49
Statistical Analysis 1: Comparison: Esomeprazole+Amox+Levo vs Esomeprazole+Bismuth+Tetra+Levo; Test type: Superiority; p < 0.001, Chi-squared

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Esomeprazole+Amox+Levo | Esomeprazole+Bismuth+Tetra+Levo
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/50
Other Adverse Events (participants affected / at risk) | 6/52 | 11/50
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Esomeprazole+Amox+Levo (N=52) | Esomeprazole+Bismuth+Tetra+Levo (N=50)
Nausea (Gastrointestinal disorders) | 4 (4) | 8 (8)
Dizziness (Gastrointestinal disorders) | 2 (2) | 3 (3)

LIMITATIONS AND CAVEATS:
The trial was performed in a single country

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-30): https://cdn.clinicaltrials.gov/large-docs/57/NCT02978157/Prot_SAP_000.pdf